CLINICAL TRIAL: NCT04038450
Title: Accuracy of Visual Range of Motion Estimates Among Physical Therapists and Physical Therapy Students
Brief Title: Accuracy of Visual Range of Motion Estimates
Status: Completed | Type: Observational
Sponsor: Methodist University, North Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 2018 - 19 0048
Record Dates: First submitted 2019-05-14; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Accuracy of Estimation of Joint Range of Motion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Practicing Physical Therapists: licensed physical therapists currently practicing
  Interventions: Other: No intervention
- Student Physical Therapists: students currently enrolled in DPT program
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No interventions separated the groups. Each group reviewed pictures and wrote down their estimated ROM of the joint pictured.

SUMMARY:
Examine the accuracy of visual estimates of various joint angles by physical therapists at various levels of education and clinical practice, taking into account years of experience, areas of practices and specialty certifications.

DETAILED DESCRIPTION:
Physical therapists oftentimes will estimate rather than measure joint range of motion. The accuracy of visual estimates of various joint measurements has not been previously assessed. No comparison has been done for years of experience and accuracy of estimations. This study will create a survey with pictures of joints at previously measured angles and therapists and students will be asked to estimate the range of motion. Various statistical analyses will be performed to determine accuracy and comparisons.

ELIGIBILITY:
Inclusion Criteria:

* licensed physical therapists
* students currently enrolled in an accredited doctorate of physical therapy program

Exclusion Criteria:

* students have not been trained in range of motion measurements
* are not licensed physical therapists

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: adults who are currently enrolled in a DPT program or graduates and licensed physical therapy practioners.
Sampling Method: Non-Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Comparison of estimated ROM to actual ROM | 6 months after completion of survey
  Compare the estimated ROM provided by the student/clinician to the actual measured ROM of the joint of the model.

CONTACTS AND LOCATIONS:
Overall Officials: Penny Schulken, DPT, Principal Investigator — Methodist University
Locations (1):
- Methodist University, North Carolina, Fayetteville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No